CLINICAL TRIAL: NCT05792046
Title: IMOvifa Perimeter Reference Database
Status: Completed | Type: Observational
Sponsor: New View Optometric Center (Industry)
Responsible Party: Sponsor
Other Study IDs: NVOC-2023-02
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Normal Eyes
MeSH Terms: interventions — Visual Field Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal: Subjects with normal visual function
  Interventions: Device: Visual field

INTERVENTIONS:
Device: Visual field — test for detecting loss in visual function

SUMMARY:
This study will collect data to establish a reference database for the IMOvifa perimeter.

DETAILED DESCRIPTION:
This study will collect data from a reference population to be used as inputs to the calculation of age corrected significance limits for expected visual function sensitivity to establish reference limits for key output parameters for select test patterns of the IMOvifa perimeter device.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older on the date of informed consent
* Able to understand the written informed consent and willing to participate
* IOP ≤ 21 mmHg (each eye)
* BCVA 20/40 or better (each eye)
* Both eyes free of ocular conditions that may affect visual function (at doctor's discretion)

Exclusion Criteria:

* Unable to tolerate ophthalmic imaging and/or VF testing
* History of conditions known to adversely affect visual function (at doctor discretion)
* Spherical Equivalent refractive error outside the range from +6 Diopters
* Cylindrical refractive error outside the range +2.5 Diopters

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with normal visual function
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Reference limit for mean deviation | Day 1
  Visual sensitivity level in decibels

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Topcon Healthcare Innovation Center, La Jolla, California
  - New View Optometric Center, La Mesa, California
  - Illinois College of Optometry, Chicago, Illinois
  - New England College of Optometry, Boston, Massachusetts